CLINICAL TRIAL: NCT01836939
Title: A Randomized Open-label Two-arm Pilot Study to Assess the Safety and Efficacy of Trichuris Suis Ova for the Treatment of Moderate to Severe Chronic Plaque Psoriasis. Protocol: Psoriasis IIT
Brief Title: Safety and Effectiveness of CNDO 201Trichuris Suis Ova (TSO) for the Treatment of Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mark Lebwohl (Other)
Collaborators: Coronado Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mark Lebwohl, Professor & Chair, Dermatology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1881
Record Dates: First submitted 2013-03-26; First posted 2013-04-22 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Psoriasis
Keywords: psoriasis, oral therapy; ova; Trichuris suis ova; TSO; CNDO 201 Trichuris suis ova
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TSO 2500 (Active Comparator): TSO 2500: 2500 embryonated, viable TSO/15 mL/day every 2 weeks X 10 weeks
  Interventions: Drug: TSO 2500
- TSO 7500 (Active Comparator): TSO 7500: 7500 embryonated, viable TSO/15 mL/day every 2 weeks X 10 weeks
  Interventions: Drug: TSO 7500

INTERVENTIONS:
Drug: TSO 2500 — TSO 2500: 2500 embryonated, viable TSO/15 mL/day every 2 weeks X 10 weeks
  Arms: TSO 2500
Drug: TSO 7500 — 12 weeks of treatment with TSO 2500 ova or TSO 7500 ova given every 2 weeks (a total of 6 doses).
  Other Names: CNDO 201 Trichuris suis ova (TSO); Trichuris suis ova; TSO; CNDO 201 Trichuris suis ova
  Arms: TSO 7500

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CNDO 201Trichuris suis ova (TSO) for the treatment of moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of CNDO 201Trichuris suis ova (TSO) for the treatment of moderate to severe plaque psoriasis.

Psoriasis is driven by T-cell infiltration in the epidermis. The T-cells involved in psoriasis exhibit a Th17-like and a Th1-like cytokine secretion profile. This excess Th17/Th1 response is thought to play a critical role in the development of psoriasis, and reducing Th17/Th1 activity would be a potential way of halting the inflammatory process leading to psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 75 years old.
* Diagnosis of stable plaque type psoriasis for at least 6 months prior to baseline
* Baseline moderate to severe psoriasis, defined as both of the following:

  1. Psoriasis covering a body surface area (BSA) ≥ 10%, and;
  2. PGA ≥ 3, and;
  3. PASI ≥ 12
* Must be in good health (except for psoriasis and psoriatic arthritis) as judged by the Investigator, based on medical history, physical examination, and clinical laboratories
* In the opinion of the investigator, must be a candidate for systemic therapy or phototherapy of psoriasis
* If a woman, before entry she must be:

  1. Postmenopausal, defined as 45 years of age with amenorrhea for at least 18 months, or > 45 years of age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level > 40 IU/mL, or Surgically postmenopausal (bilateral oophorectomy), or
  2. Surgically sterile (have had a hysterectomy or tubal ligation or otherwise be incapable of pregnancy), or
  3. If heterosexually active, practicing a highly effective method of birth control, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (eg, condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel), or male partner sterilization, consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials, for the duration of their participation in the study and for 2 months after receiving the last administration of any study agent, or
  4. Not heterosexually active
* Women of childbearing potential must have a negative pregnancy test (urine and serum) prior to randomization
* Agree to avoid prolonged exposure to natural sunlight or tanning beds or phototherapy devices for the duration of the study
* Agree to avoid any prohibited concomitant medications as detailed below for the duration of the study and for 4 weeks prior to baseline unless indication otherwise
* Negative stool culture.
* Patient has the ability to provide informed consent.

Exclusion Criteria:

* Patients with known history of intestinal parasitic infection, even if adequately treated, in the past 5 years.
* Patient received antibiotic, antifungal or antiparasitic medication in the last 2 weeks prior to Screening and/or would potentially require this during the study treatment period.
* Patient with history of drug or alcohol abuse within 6 months prior to Screening.
* Patient with evidence of poor compliance with medical advice and instruction including diet or medication.
* Patient is unable or unwilling to swallow study medication suspension.
* Patient with a significant medical condition which puts the patient at risk for study participation and/or for any reason is considered by the Investigator to be an unsuitable candidate to receive TSO or is potentially put at risk by study procedures.
* Patients who has participated in another clinical trial within 30 days of Screening for this trial and/or any experimental treatment for this population.
* White blood cell count ≤ 3,000/mm3 (≤ 3.0 x 109/L) or ≥ 14,000/mm3 (≥14 x 109/L)
* Platelet count ≤ 100,000/μL (≤100 x 109/L)
* Serum creatinine >2 x upper limit of normal (ULN)
* AST (SGOT) or ALT (SGPT) > 2 x ULN
* Total bilirubin >2 mg/dL (34 μmol/L)
* Hemoglobin < 9 g/dL
* Patients who are currently taking or have taken in the past 30 days, for any reason, any medication that, in the opinion of the investigator, suppressed the immune response. This may include but is not limited to systemic steroids, azathioprine, cyclosporine, FK506, mycophenolate mofetil, mycophenolic acid, etanercept, adalimumab, infliximab, ustekinumab, cimzia, or any other biologic agent targeted to any cell or cytokine in the immune system.
* Patients who are refractory to 2 or more biological agent plaque psoriasis therapies due to lack of efficacy.
* Patients currently taking or who have taken in the past 2 weeks, topical steroids.
* Patients on a non-stable dose of vitamin D analog in the past 30 days.
* Patients currently taking or who have taken in the past 30 days any medications likely to improve psoriasis and thus interfere with evaluation. This may include, in addition to the medications listed above, phototherapy, methotrexate, hydroxyurea, or acitretin.
* Patients with a diagnosis of inflammatory bowel disease (ulcerative colitis or Crohn's disease) or of irritable bowel syndrome
* Patients with HIV-1/HIV-2 antibody, hepatitis B surface antigen, hepatitis C antibody.
* Patient received non-steroidal anti-inflammatory drugs (NSAIDS) within 2 weeks before Baseline visit for more than 3 consecutive days, except acetylsalicylic acid ≤ 350 mg/d which is allowed.
* Women who are pregnant, intending to become pregnant, breastfeeding or planning to breastfeed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | up to 12 weeks
  The PASI score will be calculated within each patient at each protocol-specified time point. Changes and percent changes from pretreatment to each on-treatment time point will then be derived. Mean percent change from pre-treatment to Week 12.

SECONDARY OUTCOMES:
psoriasis severity | week 4
  Percentage of patients who experience an improvement in disease severity as defined by a 50%, 75%, and 90% reduction of psoriasis severity (PASI 50, PASI 75, and PASI 90 response, respectively).
psoriasis severity | week 8
  Percentage of patients who experience an improvement in disease severity as defined by a 50%, 75%, and 90% reduction of psoriasis severity (PASI 50, PASI 75, and PASI 90 response, respectively).
psoriasis severity | week 12
  Percentage of patients who experience an improvement in disease severity as defined by a 50%, 75%, and 90% reduction of psoriasis severity (PASI 50, PASI 75, and PASI 90 response, respectively).
Physicians Global Assessment (PGA) | week 4
  Percentage of patients with plaque type psoriasis who experience an improvement in disease severity as defined by a PGA ≤ 1.
Physicians Global Assessment (PGA) | week 8
  Percentage of patients with plaque type psoriasis who experience an improvement in disease severity as defined by a PGA ≤ 1.
Physicians Global Assessment (PGA) | week 12
  Percentage of patients with plaque type psoriasis who experience an improvement in disease severity as defined by a PGA ≤ 1.
Change in Body surface area (BSA) | baseline and week 12
  Body surface area (BSA) mean and percent change from pre-treatment
Change in Dermatology Life Quality Index (DLQI) | baseline and at week 12
  DLQI mean (and percent) change from pre-treatment to Week 12
safety of TSO | up to week 38
  The safety and tolerability of TSO will be evaluated via the frequency and severity of adverse events, changes in physical examinations, stool cultures, clinical laboratories, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Barrett JC, Hansoul S, Nicolae DL, Cho JH, Duerr RH, Rioux JD, Brant SR, Silverberg MS, Taylor KD, Barmada MM, Bitton A, Dassopoulos T, Datta LW, Green T, Griffiths AM, Kistner EO, Murtha MT, Regueiro MD, Rotter JI, Schumm LP, Steinhart AH, Targan SR, Xavier RJ; NIDDK IBD Genetics Consortium; Libioulle C, Sandor C, Lathrop M, Belaiche J, Dewit O, Gut I, Heath S, Laukens D, Mni M, Rutgeerts P, Van Gossum A, Zelenika D, Franchimont D, Hugot JP, de Vos M, Vermeire S, Louis E; Belgian-French IBD Consortium; Wellcome Trust Case Control Consortium; Cardon LR, Anderson CA, Drummond H, Nimmo E, Ahmad T, Prescott NJ, Onnie CM, Fisher SA, Marchini J, Ghori J, Bumpstead S, Gwilliam R, Tremelling M, Deloukas P, Mansfield J, Jewell D, Satsangi J, Mathew CG, Parkes M, Georges M, Daly MJ. Genome-wide association defines more than 30 distinct susceptibility loci for Crohn's disease. Nat Genet. 2008 Aug;40(8):955-62. doi: 10.1038/ng.175. Epub 2008 Jun 29. PMID 18587394
- [Background] Baumgart DC, Sandborn WJ. Inflammatory bowel disease: clinical aspects and established and evolving therapies. Lancet. 2007 May 12;369(9573):1641-57. doi: 10.1016/S0140-6736(07)60751-X. PMID 17499606
- [Background] Crohn BB, Ginzburg L, Oppenheimer GD. Regional ileitis: a pathologic and clinical entity. 1932. Mt Sinai J Med. 2000 May;67(3):263-8. No abstract available. PMID 10828911
- [Background] Loftus EV Jr, Schoenfeld P, Sandborn WJ. The epidemiology and natural history of Crohn's disease in population-based patient cohorts from North America: a systematic review. Aliment Pharmacol Ther. 2002 Jan;16(1):51-60. doi: 10.1046/j.1365-2036.2002.01140.x. PMID 11856078